CLINICAL TRIAL: NCT02122081
Title: A Feasibility Study of Organ-Sparing Marrow-Targeted Irradiation (OSMI) to Condition Patients With High-Risk Hematologic Malignancies Prior to Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Organ-Sparing Marrow-Targeted Irradiation Before Stem Cell Transplant in Treating Patients With High-Risk Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumithira Vasu (Other)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13219; NCI-2014-00763 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Radiotherapy; Radiation; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Methotrexate; merphos; Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (OSMI, allogeneic transplant) (Experimental): CONDITIONING REGIMEN: Patients undergo organ-sparing marrow irradiation BID on days -6 to -4 and receive cyclophosphamide IV over 1-2 hours every 24 hours on days -3 to -2. Patients with an unrelated donor also receive anti-thymocyte globulin every 24 hours on days -4 to -2.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 and continuing for at least 6 months and methotrexate IV on days 1, 3, 6, and 11.
  TRANSPLANT: Patients undergo allogeneic peripheral blood progenitor cell or bone marrow transplant on day 0.
  Interventions: Radiation: radiation therapy; Drug: cyclophosphamide; Biological: anti-thymocyte globulin; Drug: tacrolimus; Drug: methotrexate; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: radiation therapy — Undergo organ-sparing marrow irradiation BID on days -6 to -4
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: cyclophosphamide — Given IV over 1-2 hours every 24 hours on days -3 to -2.
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: anti-thymocyte globulin
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic peripheral blood progenitor cell or bone marrow transplant on day 0
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic peripheral blood progenitor cell or bone marrow transplant
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic peripheral blood progenitor cell or bone marrow transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial aims to assess feasibility and tolerability of using an LINAC based "organ-sparing marrow-targeted irradiation" to condition patients with high-risk hematological malignancies who are otherwise ineligible to undergo myeloablative Total body irradiation (TBI)-based conditioning prior to allogeneic stem cell transplant. The target patient populations are those with ALL, AML, MDS who are either elderly (>50 years of age) but healthy, or younger patients with worse medical comorbidities (HCT-Specific Comorbidity Index Score (HCT-CI) > 4). The goal is to have the patients benefit from potentially more efficacious myeloablative radiation based conditioning approach without the side effects associated with TBI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility and tolerability of OSMI based hematopoietic stem cell transplant (HSCT) as defined by transplant-related mortality (TRM) at day 30 as well as rate of grade II/III organ toxicity (defined by Bearman Regimen-Related Toxicities Scale) attributable to conditioning occurring within 30 days.

SECONDARY OBJECTIVES:

I. Day 100 transplant-related mortality (TRM). II. Donor chimerism assessment at day 100 (to assess failure of engraftment rate).

III. Incidence of acute graft-versus-host disease (aGVHD) by day 100. IV. Incidence of chronic GVHD at one year. V. Cumulative incidence of grade II organ toxicity through day 100. VI. Rate and kinetics of hematopoietic recovery. VII. Incidence of graft failure (primary and secondary). VIII. Rate of infectious complications. IX. Cumulative incidence of relapse, overall survival, and progression-free survival at 1 year.

OUTLINE:

CONDITIONING REGIMEN: Patients undergo organ-sparing marrow irradiation twice daily (BID) on days -6 to -4 and receive cyclophosphamide intravenously (IV) over 1-2 hours every 24 hours on days -3 to -2. Patients with an unrelated donor also receive anti-thymocyte globulin every 24 hours on days -4 to -2.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV or orally (PO) beginning on day -1 and continuing for at least 6 months and methotrexate IV on days 1, 3, 6, and 11.

TRANSPLANT: Patients undergo allogeneic peripheral blood progenitor cell or bone marrow transplant on day 0.

After completion of study treatment, patients are followed up weekly for 12 weeks, at day 100, and then at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or myelodysplastic syndromes (MDS) with fewer than 10% myeloblasts or lymphoblasts in the bone marrow and no blasts in the peripheral blood on morphologic analysis performed within 30 days of start of the conditioning regimen; if remission bone marrow is available beyond 30 days a new bone marrow evaluation is required to assess remission status

  * The diagnosis of AML, ALL, or MDS will be based on World Health Organization (WHO) criteria
  * Pre-transplant bone marrow sample must be evaluable for assessment of remission status (i.e. aspirate smear containing particles and/or evaluable bone marrow core biopsy)
  * Patients with leukemia infiltration in the central nervous system (CNS) are eligible if cerebrospinal fluid (CSF) cytospin is negative for myeloblasts or lymphoblasts at time of enrollment
  * If the patient has an intra-abdominal chloroma on presentation, and has a partial response or complete response to treatment (size reduction of chloroma and marrow blast < 10%), the patient is eligible; however the chloroma must be included as part of the treatment target
* For patients receiving treatment of their AML, MDS or ALL prior to transplantation:

  * Interval between the start of a cycle of conventional cytotoxic chemotherapy and the start of conditioning regimen must be at least 30 days
  * Interval between completing treatment with a hypomethylating agent or other non-cytotoxic chemotherapy and the start of conditioning regimen must be at least 10 days
* Hematopoietic Cell Transplantation-Specific Comorbidity Index score (HCT-CI) =< 4 for patients in Cohort 1 and > 4 for Cohort 2
* Patient must be able to lie still in full body cast for 45 minutes
* Must have a suitable donor defined as a sibling matched at 5/6 or 6/6 antigens (human leukocyte antigen [HLA]-A, B, and DRB1) or an unrelated volunteer matched at 7/8 or 8/8 HLA alleles (HLA-A, B, C, and DRB1)
* Signed informed consent
* DONOR: "High resolution" typing at HLA-A, B, C and DRB1 alleles

  * Single antigen mismatch for siblings and single allele mismatch for volunteer unrelated donors is acceptable
  * Donors must be >= 17 years of age

Exclusion Criteria:

* Circulating peripheral blood myeloblasts or lymphoblasts on morphologic analysis from time of last treatment to time of enrollment
* Prior allograft or prior autograft
* Active CNS disease as identified by positive CSF cytospin at time of enrollment
* Karnofsky performance score < 70
* Symptomatic uncontrolled coronary artery disease or ejection fraction < 40%
* Total bilirubin >= 2 x the upper limit of normal
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >= 3 x the upper limit of normal
* Diffusion capacity of the lung for carbon monoxide (DLCO) < 40%
* Forced expiratory volume in one second (FEV1) < 50% (corrected for hemoglobin)
* Receiving supplementary continuous oxygen
* Creatinine clearance < 50 mL/min/1.73m^2
* Patients with active uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms)
* Patients seropositive for the human immunodeficiency virus (HIV)
* Females who are pregnant or breastfeeding
* Fertile men and women unwilling to use contraceptive techniques during and for 12 months following treatment
* Patients who had prior radiation to more than 20% bone marrow containing areas or to any areas exceeding 2000 cGy
* DONOR:

  * Donors will be excluded if they are an identical twin of the recipient
  * Females who are pregnant (positive serum beta human chorionic gonadotropin beta [β HCG]) or uninterruptible breastfeeding
  * HIV seropositive
  * Donors receiving experimental therapy or investigational agents unless approved by the protocol chair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
TRM, defined as death occurring in a patient from causes other than disease relapse | At day 30 post-transplant
  Proportions will be derived for incidence of TRM divided by all evaluable patients along with corresponding 95% binomial confidence intervals.
Rate of grade II/III organ toxicity, defined by the Bearman Regimen-Related Toxicities Scale | Up to 30 days
  Toxicities will be tabulated by grade for each cohort, by type of toxicity, as well as the maximum grade overall. Toxicity frequencies will be described for the day +30, day +100, and one year time intervals as well as cumulative over time. Proportions will be derived for incidence of grade II/III organ toxicity divided by all evaluable patients along with corresponding 95% binomial confidence intervals.

SECONDARY OUTCOMES:
TRM | Day 100 post-transplant
  Proportions will be derived for incidence of toxicity divided by all evaluable patients along with corresponding 95% binomial confidence intervals.
Donor chimerism | Day 100
  Donor chimerism is used to assess failure of engraftment rate.
Incidence of aGVHD, graded according to Ohio State University Bone Marrow Transplant (OSU BMT) Program policy | Up to day 100
  The first day of aGVHD onset at a certain grade will be used to calculate cumulative incidence curves for that GVHD grade.
Incidence of chronic GVHD, scored according to the OSU BMT Program policy | At 1 year
  The first day of chronic GVHD onset will be used to calculate cumulative incidence curves. Rates and severity of chronic GHVD will be calculated.
Cumulative incidence of grade II organ toxicity | Up to day 100
  Toxicity will be tabulated by grade for each cohort, by type of toxicity as well as the maximum grade overall.
Incidence of hematopoietic recovery | Up to day 100
  The rate and kinetics of hematopoietic recovery will be assessed. The kinetics of post-transplant recovery of both neutrophil and platelet engraftment will be assessed.
Incidence of graft failure | Up to 1 year post-transplant
  Primary graft failure (defined by the lack of neutrophil engraftment by 28 days) and secondary graft failure (defined by initial neutrophil engraftment followed by subsequent decline in neutrophil counts < 500/uL unresponsive to growth factor therapy) will be assessed on days 30 and 100 and at 1 year post-transplant.
Rate of infectious complications | Up to 12 months
  The number of infections and the number of patients experiencing infections will be tabulated by type of infection, severity, and time period after transplant. The cumulative incidence of severe, life-threatening, or fatal infections will be tabulated.
Incidence of relapse | Time from start of conditioning to relapse, assessed at 1 year
Overall survival | Time from start of conditioning to death, loss to follow up, or end of study, whichever comes first, assessed at 1 year
Progression-free survival | Time from start of conditioning to relapse, progression, death, initiation of non-protocol therapy, loss to follow up or end of study, whichever comes first, assessed at 1 year
  Patients are considered a failure of this endpoint if they die or suffer from disease relapse or progression.
Immune reconstitution | Up to 12 months post transplant
  Quantitative assessments of peripheral blood CD3, CD4, CD8, CD19, and CD56 positive lymphocytes will be done throw flow cytometric analysis at baseline, 100 days, and 12 months post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu